CLINICAL TRIAL: NCT00639795
Title: Prospective Randomized Trial Evaluating the Effects of Paravertebral Nerve Blocks on Postoperative Pain and the Perioperative Inflammatory Response Following Video Assisted Thorascopic Surgery
Brief Title: Study of the Effect of Regional Nerve Blocks on Pain and Inflammation After Video Assisted Thorascopic Lung Surgery
Acronym: VATS_IM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate sample population
Sponsor: Memorial Medical Center (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: William T Fritz, M.D., Laurel Anesthesia Group, Memorial Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A-13101.2 MMC 06-28; Proposal Log Number 04070001; Award Number W81XWH-05-1-0047
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Pain
Keywords: Thoracic paravertebral block; Cytokines; Video assisted thorascopic surgery; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients randomized to receive thoracic paravertebral nerve blockade in addition to general endotracheal anesthesia during video assisted thoracoscopy procedure
  Interventions: Procedure: Thoracic Paravertebral Nerve Block
- B (Sham Comparator): Patients randomized to receive sham single-injection thoracic peripheral nerve blockade (no injection) in addition to general endotracheal anesthesia
  Interventions: Procedure: Thoracic Paravertebral Nerve Block

INTERVENTIONS:
Procedure: Thoracic Paravertebral Nerve Block — One Single-injection, thoracic peripheral nerve blockade performed intraoperatively following patient induction with general endotracheal anesthesia
  Other Names: VATS IM; Thoracic Peripheral Nerve Blockade
  Arms: A
Procedure: Thoracic Paravertebral Nerve Block — Sham single-injection thoracic peripheral nerve blockade following patient induction with general endotracheal anesthesia
  Arms: B

SUMMARY:
The purpose of this study is to compare:

1. The degree of systemic postoperative inflammation (cytokine measurement) with the degree of post-operative pain
2. The degree of pain and nausea and
3. The pre and post operative pulmonary functions

following Video Assisted Thorascopic Surgery (VATS) performed under general anesthesia with the addition of intra-operative single-injection paravertebral blockade vs general anesthesia with a sham intra-operative paravertebral nerve blockade

DETAILED DESCRIPTION:
* Enrolled subjects scheduled to undergo video-assisted thorascopic surgery (VATS) will be randomized to receive either paravertebral block or placebo(adhesive bandage applied at the site).
* All patients will undergo a standardized general anesthetic regimen.
* Human biological specimens will be collected preoperatively, postoperatively (in the PACU) at the first morning blood draw of POD 1, POD 2, POD 3, and POD 10-14 (follow-up visit at surgeons office)and analyzed for CRP, Cortisol & inflammatory markers (IL-1beta,IL-2,IL-4,IL-5,IL-6, IL-8, IL-10,INF-gamma, TNF-alpha)
* Pulmonary functions (FEV1/FEV6) will be performed in the pre-op holding area prior to sedation and post-operatively on the morning of post-op day 1.
* Pain levels will be assessed with the Wong-Baker Faces and Visual Analog Scale pre-operatively in the PACU and hourly for a total of 6 hours and then every 8 hrs.and with patient self-report in diary after discharge.
* Pain levels will be assessed with the McGill-Melzack Pain Questionnaire pre-operatively, the evening of POD1-POD3 and by patient self-report in diary after discharge.
* Nausea assessments will occur at arrival on floor and every 8 hours thereafter until discharge.
* Narcotic requirements will be collected daily in the hospital and by patient self report in diary thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Planned thoracoscopy with low probability(by surgeon estimate) of conversion to open procedure

Exclusion Criteria:

* Age less than 18
* Clinical or laboratory evidence of systemic infection
* Current pregnancy as assessed by preoperative urine HCG test
* Serious, uncontrolled, non-malignant illness
* Malignant illness requiring systemic chemotherapy in the last 6 months
* Documented allergy to oxycodone, morphine sulfate or acetaminophen
* Contraindication to peripheral nerve blockade or general anesthesia including:

  1. patient refusal
  2. active infection at site of planned block
  3. documented allergy to any local or general anesthetic medications
  4. significant coagulopathy( prothrombin time >15 seconds, INR>1.5
  5. pre-existing neuropathy and medical conditions or deformities which would compromise block or anesthetic safety
* Planned pleurodesis
* Current use of high dose inhaled or systemic steroids
* Current use of Amiodarone (Cordarone)
* Morbid obesity (BMI=40kg/m2)
* Patients with clinically significant mental health issues such as psychosis requiring treatment with antipsychotic medications.
* Patients unable to consent
* Patients with active infections requiring antibiotics within one month of registration
* Participation in other clinical trials that may interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Comparing the degree of systemic post-operative inflammation with the degree of post-operative pain | 1 year

SECONDARY OUTCOMES:
To compare the degree of pain and nausea | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William T Fritz, MD, Principal Investigator — Memorial Medical Center
Locations (1):
- Memorial Medical Center, Johnstown, Pennsylvania, United States